CLINICAL TRIAL: NCT03027232
Title: Control of Leukocyte Function
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Wolfgang Junger, Professor of Surgery, Beth Israel Deaconess Medical Center
Other Study IDs: 2007P000215
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Inflammation, Brain
Keywords: infection
MeSH Terms: conditions — Encephalitis; Infections | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood is collected from all subjects in the same fashion. Purpose: isolation of immune cells for in vitro studies of cell function.
  This is an observational study in human beings in predefined groups of individuals who are healthy and volunteer to donate blood for laboratory science studies. Subjects in the study receive neither diagnostic, therapeutic, nor other interventions, and the investigator does not assign specific interventions to any of the subjects of the study.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention (drugs) will be given. Purpose: collecting blood for in vitro studies — No drugs or interventions are given. Single purpose is to draw blood from healthy subjects to study immune cell biology in vitro. No records about subjects to be kept.

SUMMARY:
The protocol is to draw peripheral blood from healthy volunteers for in vitro studies. The aims of these in vitro studies are to determine the cellular and intracellular mechanisms by which hypertonic saline and ATP release regulate neutrophil and lymphocyte functions.

DETAILED DESCRIPTION:
The proper regulation of leukocyte function is critical for immune defense and to prevent autoimmune diseases. Many aspects of immune cell regulation are unknown. A better understanding could lead to novel therapeutic approaches to improve immune function in patients suffering from various diseases.

The investigators have found that hypertonic conditions regulate leukocyte functions through feedback mechanisms involving ATP release and purinergic receptors. The purpose of the proposed protocol is to obtain access to peripheral blood from healthy volunteers to study these complex regulatory mechanisms in more detail.

ELIGIBILITY:
Inclusion Criteria:

* any healthy volunteer

Exclusion Criteria:

* pregnancy
* needing/using drugs
* inflammatory or infectious complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Immune cells will be studied in vitro to learn about basic mechanisms of immune cell signaling. | Blood is collected as needed; time frame: indefinitely. Blood used between 1-7 days after blood draws.
  The purpose of this study is to obtain blood from healthy subjects (volunteers) for in vitro studies to explore how immune cells function. Cells will be isolated and subjected to various tests including stimuli that simulate immune cell activation in health and disease. Subjects will not be subjected to any treatments. Only some of the cells (leukocytes) in the blood will be studied. For example, activation events such as cytokine production, the ability of leukocytes (=immune cells) to detect and respond to bacterial products will be assessed. No identifiable information about study subjects will be kept.

CONTACTS AND LOCATIONS:
Locations (1):
- BIDMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No